CLINICAL TRIAL: NCT01507350
Title: Effects of Obesity Surgery on Renal Function
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Carel Le Roux, Consultant metabolic medicine, Imperial College London
Other Study IDs: BSR
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Impaired Renal Function
Keywords: obesity related glmerulopathy; 51 Cr-EDTA clearance; impaired renal function; gastric band; GFR measurement; gastric bypass; sleeve gastrectomy
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obesity Surgery: Patients having gastric band, sleeve gastrectomy, and gastric bypass will have blood and urine tests, and 51 Cr-EDTA clearance to assess renal function. These are taken before and after the surgery at 6 weeks , 6 months and 12 months.

SUMMARY:
Increasing risk of impaired renal function as a result of obesity is well known. Early data has postulated that weight loss might improve kidney function, but the evidence is rather limited due to the difficulties in measuring glomerular filtration rate(GFR) after weight loss. Cystatin C, GFR measurement using Cockcroft-Gault (CCG) and Modification of Diet in Renal Disease (MDRD) equations, have all yield conflicting results after weight loss surgery.

The study aim to assess:

1. use of 51Cr-EDTA Clearance as the methodological gold standard in evaluating changes in renal function before and after weight loss surgery.
2. the reliability of using MDRD, CCG and Cystatin C in measuring GFR after weight loss surgery
3. the differences in alterations in renal function dependent on the surgical procedures( gastric bypass, gastric band, sleeve gastrectomy).
4. the use of urine albumin/creatinine ratio in detecting alterations in microalbuminuria.

DETAILED DESCRIPTION:
This is a prospective study on obese human subjects undergoing bariatric surgery. Forty-five patients due to undergo gastric bypass (n=15), gastric banding (n=15), and gastric sleeve surgery (n=15) will be recruited.

Subjects will be screened prior to entry into the study with full history, examination, routine bloods (FBC, U+E, liver function tests, and glucose).

1. Blood samples and 24h urine specimens are taken at four time points: preoperatively as well 6 weeks, 6 and 12 months postoperatively.
2. The following methods of GFR assessment will be executed the same time point: measurement of serum creatinine concentration, calculation of the abbreviated and extended MDRD formulae, CCG, creatinine clearance, serum Cystatin C concentration and the 51Chromium-EDTA clearance.

Inclusion criteria

1. Patients with a BMI of >35kg/m2 approved for obesity surgery based on the NICE criteria.
2. Patients with a GFR <60 mL/min/1.73

Exclusion criteria

1. Allergy to chromium

ELIGIBILITY:
Inclusion Criteria:

* Patients with a BMI of >35kg/m2 approved for obesity surgery based on the NICE criteria.
* Patients with a GFR <60 mL/min/1.73 m2

Exclusion Criteria:

* Allergy to chromium

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with a BMI of >35kg/m2 approved for obesity surgery based on the NICE criteria.
  2. Patients with a GFR <60 mL/min/1.73 m2
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2011-06; Primary Completion 2016-06-01 (Actual); Study Completion 2016-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carel W le Roux, MBChB, PhD, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chuah LL, Miras AD, Perry LM, Frankel AH, Towey DJ, Al-Mayahi Z, Svensson W, le Roux CW. Measurement of glomerular filtration rate in patients undergoing obesity surgery. BMC Nephrol. 2018 Dec 29;19(1):383. doi: 10.1186/s12882-018-1188-7. PMID 30594245

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obesity Surgery
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Obesity Surgery
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 62.0 [50.5 to 63.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
BMI (kg/m^2) [Mean (Full Range); unit: kg/m^2] | 45.5 [42.2 to 47.8]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Glomerular Renal Function After Weight Loss Surgery as Measured by 51Cr-EDTA Clearance
Description: The outcome measure is reported as the number of participants who achieved a change in the glomerular renal function after weight loss surgery as measured by 51Cr-EDTA Clearance.
  51Cr-EDTA GFR was ascertained using bolus injection of 1.46-2.66 MBq 51Cr-EDTA, with between 6 and 8 venous blood samples were collected at approximately 15, 30, 60, 90, 120, 180, 240, and 300 min to assess 51Cr-EDTA clearance. 51Cr-EDTA GFR was calculated using the Bi-exponential Fitting Method described in the British Nuclear Medicine Society guidelines. The prepared standard and patient samples were counted for 15 and 60 mins respectively using a Wallac 1470 Wizard Gamma Counter (Perkin Elmer Inc., Waltham, Massachusetts, USA). The measured GFR was scaled to BSA in order to maintain uniformity in comparison to reported eGFR.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Obesity Surgery
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: No difference
Arm/Group | Obesity Surgery
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes